CLINICAL TRIAL: NCT00601172
Title: A Study of Single Dose Intravenous Casopitant in Combination With Ondansetron and Dexamethasone for the Prevention of Oxaliplatin Induced Nausea and Vomiting.
Brief Title: A Study Of IV Casopitant For The Prevention Of Chemotherapy Induced Nausea And Vomiting.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NKV110721
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-11

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: vomiting; colorectal cancer; nausea; oxaliplatin
MeSH Terms: conditions — Nausea; Vomiting; Colorectal Neoplasms | interventions — casopitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Placebo + standard antiemetics
  Interventions: Drug: Dexamethasone; Drug: Placebo; Drug: Ondansetron
- Single Dose IV (Experimental): Casopitant + standard antiemetics
  Interventions: Drug: Casopitant; Drug: Dexamethasone; Drug: Ondansetron

INTERVENTIONS:
Drug: Casopitant — Experimental NK-1 receptor antagonist
  Arms: Single Dose IV
Drug: Dexamethasone — Standard antiemetics
Drug: Placebo — Placebo to match IV casopitant
  Arms: Control
Drug: Ondansetron — Standard antiemetics

SUMMARY:
This a Phase III trial designed to determine if IV casopitant plus dexamethasone and ondansetron is more effective in the prevention of vomiting and nausea then dexamethasone and ondansetrone alone following the administration of moderately emetogenic oxaliplatin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be considered eligible for initial inclusion in this study, and progression into subsequent cycles of therapy within the study, only if all of the following criteria apply:
* Subject understands the nature and purpose of this study and the study procedures and has signed an informed consent form for this study to indicate this understanding.
* At least 18 years of age.
* Is scheduled to receive oxaliplatin at a dose between 85 mg/m² and 130 mg/m² in their first cycle of therapy for the treatment of colorectal cancer, administered as a single IV dose over 2-6 hours on Day 1 only, in combination with 5FU/LV, or in combination with capecitabine.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Hematologic and metabolic status adequate for receiving an oxaliplatin-based moderately emetogenic regimen and meeting the following criteria:

  * Total Neutrophils ≥1500/mm³ (Standard units : ≥1.5 x 10^9/L)
  * Platelets ≥100,000/mm³ (Standard units: ≥100.0 x 10^9/L)
  * Bilirubin ≤1.5 x upper limit of normal (ULN)
  * Serum Creatinine ≤1.5 mg/dL (Standard units : ≤132.6 µmol/L) OR
  * Creatinine clearance ≥60 mL/min

Creatinine clearance must be calculated using the Cockcroft-Gault formula:

Clcreat (ml/min) = (140-age [yr]) x body wt [kg] 72 x serum creatinine [mg/dl] For females: multiply creatinine clearance by a factor of 0.85. OR Clcreat (ml/min) = K x (140-age [yr]) x body wt [kg] serum creatinine [µmol/L] K=1.05 for females K=1.23 for males

* Liver enzymes must be below the following limits:
* Without known liver metastases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 x ULN.
* With known liver metastases: AST and/or ALT ≤5.0 x ULN.

  * Is willing and able to complete daily components of the Subject Diary for Cycle 1 and Cycle 2 without assistance from others.
  * A female subject is eligible to enter and participate in this study if she is of:

    1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses)
    2. child-bearing potential: must have a negative serum pregnancy test result or negative urine dipstick pregnancy test within 24 hours prior to the first dose of investigational product on Cycle 1 Day 1. Women of childbearing potential must also commit to consistent and correct use of an acceptable method of birth control. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject;
* oral contraceptives (e.g., oral, injectable, or implantable) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm for a period after the trial to account for a potential drug interaction (minimum of six weeks);
* double-barrier method of contraception consisting of spermicide with either condom or diaphragm;
* intra-uterine device with a documented failure rate of less than 1% per year;
* complete abstinence from intercourse for two weeks before exposure to the investigational product throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of 3 days);
* if subject indicates they will remain abstinent during the period described above, they must agree to follow GSK guidelines for the consistent and correct use of an acceptable method of birth control should they become sexually active.

Exclusion Criteria:

* A subject will not be eligible for initial inclusion in this study if any of the following criteria apply, or will not be eligible for subsequent cycles of therapy if any of the following criteria become applicable:
* Has received cytotoxic chemotherapy prior to the first study cycle of chemotherapy, with the exception that previous adjuvant therapy with 5FU/LV or capecitabine is permitted, provided that the last dose of adjuvant therapy was completed at least 6 months prior to receiving the first dose of study medication or investigational product. Previous biological or hormonal therapy completed at any time is permitted.
* Scheduled to receive chemotherapy with any cytotoxic agents (e.g., irinotecan, gemcitabine) or biological agents (e.g., cetuximab, panitumimab) other than the protocol allowed chemotherapy described in Inclusion Criterion 3.
* Is a female subject who is pregnant or lactating.
* Has received radiation therapy in the 10 days prior to the first dose of study medication or investigational product and/or is scheduled to receive such radiation therapy in the 6 days following the first dose of study medication or investigational product in the first cycle of chemotherapy. Radiation therapy may be added in subsequent cycles of chemotherapy.
* Has experienced emesis (i.e., vomiting and/or retching) or clinically significant nausea in the 24 hours preceding the first dose of study medication or investigational product for each cycle of chemotherapy.
* Has known central nervous system metastasis, unless previously successfully treated with excision or radiation, and has been stable for at least 1 week immediately prior to receiving the first dose of study medication or investigational product.
* Has increased intracranial pressure, hypercalcemia, an active systemic infection, or any uncontrolled medical condition (other than malignancy) which in the opinion of the Investigator may confound the results of the study, represent another potential etiology for emesis and nausea (other than CINV) or pose an unwarranted risk to the subject.
* Has a known hypersensitivity or contraindication to ondansetron, another 5-HT3 receptor antagonist, dexamethasone, or any component of casopitant.
* Has received an NK-1 receptor antagonist prior to the first study cycle of chemotherapy.
* Has received an investigational drug within the previous 30 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study medication or investigational product, or is scheduled to receive any investigational drug other than casopitant/placebo during the study period.
* Has taken/received any medication of moderate or high emetogenic potential (including antineoplastic agents [see Appendix 2]) within the 48 hours prior to the first dose of study medication or investigational product in each cycle. However, opioid narcotics will be permitted if the subject has been on such medication for at least 7 days at a stable dose prior to the start of each cycle, and has not experienced emesis or nausea from the narcotics.
* Has taken/received any medication with known or potential antiemetic activity within the 24-hour period (unless otherwise stated) prior to receiving the first dose of study medication or investigational product or is expected to require use of such medication during the 120 hour assessment period for Cycle 1 of therapy only. This includes, but is not limited to:

  * 5-HT3 receptor antagonists (e.g., additional ondansetron, or granisetron, dolasetron, tropisetron, ramosetron). Palonosetron is not permitted within 7 days prior to administration of study medication or investigational product;
  * benzamide / benzamide derivatives (e.g., metoclopramide, alizapride);
  * benzodiazepines (except if the subject is receiving such medication for sleep or anxiety and has been on a stable dose for at least 7 days prior to the first dose of investigational product; however, lorazepam is prohibited 24 hours prior to receiving study drug regardless of reason for use);
  * phenothiazines (e.g., prochlorperazine, promethazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine);
  * butyrophenones (e.g., haloperidol, droperidol);
  * corticosteroids within 72 hours prior to the first dose of study medication or investigational product (e.g., dexamethasone, methylprednisolone); with the exception that topical steroids for skin disorders including eye and ear drops, and inhaled steroids for respiratory disorders at ≤ 10 mg prednisone daily or its equivalent are permitted;
  * anticholinergics (e.g., scopolamine); with the exception that anticholinergics for the treatment of respiratory disorders and the management of diarrhea (e.g., ipratropium bromide, and hyoscyamine) and anticholinergic eye drops are permitted;
  * first-generation antihistamines (e.g., cyclizine, hydroxyzine, diphenhydramine; see Appendix 4); except for topical use which is permitted;
  * domperidone;
  * cannabinoids;
  * mirtazapine;
  * olanzapine.
* Has taken/received strong or moderate inhibitors of CYP3A4 and CYP3A5 for a specified period prior to administration of investigational product in each cycle of therapy.
* Has taken/received inducers of CYP3A4 and CYP3A5 within 14 days prior to the administration of investigational product in each cycle of therapy.
* Is currently taking, or plans to take the following CYP2C8 substrates at any time during the study: the anti-diabetic agent repaglinide or the diuretic torsemide.
* Is currently taking, or plans to take any of the following CYP3A4 substrates at any time during the study: astemizole, cisapride, pimozide, terfenadine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2008-03-10 (Actual); Primary Completion 2009-04-13 (Actual); Study Completion 2009-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (89):
- United States (22):
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Corona, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Hilton Head Island, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Burlington, Vermont
- Belgium (4):
  - GSK Investigational Site, Assebroek
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Ottignies
- Bulgaria (3):
  - GSK Investigational Site, Shumen
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (9):
  - GSK Investigational Site, Sault Ste. Marie, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Rimouski, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Czechia (5):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Havlíčkův Brod
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Semily
- Germany (19):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Hof, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Bad Soden, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Braunschweig, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Recklinghausen, North Rhine-Westphalia
  - GSK Investigational Site, Würselen, North Rhine-Westphalia
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Pinneberg, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Hamburg
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Veszprém
- Italy (12):
  - GSK Investigational Site, Potenza, Basilicate
  - GSK Investigational Site, Rionero in Vulture (PZ), Basilicate
  - GSK Investigational Site, Reggio Calabria, Calabria
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Terni, Umbria
  - GSK Investigational Site, Padua, Veneto
- Russia (5):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Moscow Region
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
- Slovakia (4):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Poprad
- South Korea (3):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul

REFERENCES:
- [Background] Hesketh PJ, Wright O, Rosati G, Russo M, Levin J, Lane S, Moiseyenko V, Dube P, Kopp M, Makhson A. Single-dose intravenous casopitant in combination with ondansetron and dexamethasone for the prevention of oxaliplatin-induced nausea and vomiting: a multicenter, randomized, double-blind, active-controlled, two arm, parallel group study. Support Care Cancer. 2012 Jul;20(7):1471-8. doi: 10.1007/s00520-011-1235-4. Epub 2011 Aug 7. PMID 21822913

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 89 centers (55 centers in Europe, 30 in North America and 4 in Korea) in 11 countries from 10-March-2008 to 13-April-2009.
Pre-assignment Details: All participants received ondansetron and dexamethasone as background antiemetic therapy. To assure adequate blinding, placebo to match casopitant was used. Participants were screened within 14 days of first dose of study anti-emetics and were randomly assigned to either single dose intravenous (IV) (90 mg casopitant) or control (placebo).
Groups:
- Placebo: Eligible participants received placebo to match casopitant, via IV route, (along with Ondansetron 8 milligram [mg] twice daily [BID] orally and dexamethasone 8 mg IV) on Day 1 of each cycle over 30 minutes.
- Casopitant 90 mg: Eligible participants received casopitant 90 mg, via IV route, (along with Ondansetron 8 mg BID orally and dexamethasone 8 mg IV) on Day 1 of each cycle over 30 minutes.
Period: Overall Study
Arm/Group | Placebo | Casopitant 90 mg
Started | 355 | 355
Completed | 214 | 228
Not Completed | 141 | 127
Not completed — Adverse Event | 43 | 32
Not completed — Lack of Efficacy | 11 | 12
Not completed — Protocol Violation | 2 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Physician Decision | 27 | 28
Not completed — Withdrawal by Subject | 35 | 27
Not completed — Did not meet continuation criteria | 19 | 20

BASELINE CHARACTERISTICS:
Population: For Age, only 352 participants were analyzed in the Placebo group.
Groups:
- Placebo: Eligible participants received placebo to match casopitant, via IV route, (along with Ondansetron 8 mg BID orally and dexamethasone 8 mg IV) on Day 1 of each cycle over 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Placebo | Casopitant 90 mg | Total
Number analyzed (Participants) | 355 | 355 | 710
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age data is presented for modified Intent-to-Treat (mITT) Population which comprised of all participants who were randomized, received any investigational product and had oxaliplatin administered. Population: N=352
  Years
    number analyzed (Participants) | 352 | 355 | 707
    (all) | 61.3 (10.77) | 61.3 (11.03) | 61.3 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 173 | 318
  Male | 210 | 182 | 392
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 24 | 30 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 326 | 318 | 644
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Complete Response in the Overall Phase (0-120 Hours) Following Initiation of the First Cycle of an Oxaliplatin Based Moderately Emetogenic Chemotherapy (MEC) Regimen
Description: Complete response was defined as no vomiting, no retching and no use of anti-emetic rescue medication. Participants who vomited or retched or received rescue medication in the acute phase (0- 24 hours) following administration of oxaliplatin were also considered as complete response failures in the subsequent delayed (24-120 hour) time period, irrespective of actual response in the delayed phase. However, participants who vomited or retched or received rescue medication in the delayed (24-120 hours) phase were not considered as failures in the acute (0-24 hours) phase. The overall phase began at the start of the administration of the oxaliplatin infusion. Percentage of participants who achieved a complete response in the overall phase (0-120 hours) are presented.
Time Frame: 0 to 120 hours in the first cycle of chemotherapy
Population: Modified Intent-to-Treat Population (mITT) comprised of all participants who were randomized, received any investigational product and had oxaliplatin administered.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants | 85 | 86
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg; Test type: Superiority or Other; p = 0.7273, Pooled Z test — p-value based on normal approximation to the binomial using a pooled Z test; difference in percentage of participants = 1.0, 95% CI 2-sided [-4.6 to 6.6] — The parameter estimated was difference in percentage of participants with response

2. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response in the Acute Phase of Cycle 1
Description: Complete response was defined as no vomiting, no retching and no use of anti-emetic rescue medication. Participants who vomited or retched or received rescue medication in the acute phase (0- 24 hours) following administration of oxaliplatin were also considered as complete response failures in the subsequent delayed (24-120 hour) time period, irrespective of actual response in the delayed phase. However, participants who vomited or retched or received rescue medication in the delayed (24-120 hours) phase were not considered as failures in the acute (0-24 hours) phase. Percentage of participants who achieved a complete response in the acute phase of Cycle 1 are presented.
Time Frame: 0 to 24 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants | 96 | 97
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg; Test type: Superiority or Other; p = 0.4771, Pooled Z test — p-value based on normal approximation to the binomial using a pooled Z test; Difference in percentage of participants = 1.0, 95% CI 2-sided [-1.8 to 3.8] — The parameter estimated was difference in percentage of participants with response

3. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response in the Delayed Phase of Cycle 1
Description: Complete response was defined as no vomiting, no retching and no use of anti-emetic rescue medication. Participants who vomited or retched or received rescue medication in the acute phase (0- 24 hours) following administration of oxaliplatin were also considered as complete response failures in the subsequent delayed (24-120 hour) time period, irrespective of actual response in the delayed phase. However, participants who vomited or retched or received rescue medication in the delayed (24-120 hours) phase were not considered as failures in the acute (0-24 hours) phase. Percentage of participants who achieved a complete response in the delayed phase of Cycle 1 are presented.
Time Frame: 24 to 120 hours (delayed phase) in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants | 85 | 86
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg; Test type: Superiority or Other; p = 0.7273, Pooled Z test; p-value based on normal approximation to the binomial using a pooled Z test; Difference in percentage of participants = 1.0, 95% CI 2-sided [-4.6 to 6.6] — The parameter estimated was difference in percentage of participants with response

4. Secondary Outcome: Percentage of Participants Who Achieved a Complete Response in the Overall Phase of Cycle 2
Description: Complete response was defined as no vomiting, no retching and no use of anti-emetic rescue medication. Participants who vomited or retched or received rescue medication in the acute phase (0- 24 hours) following administration of oxaliplatin were also considered as complete response failures in the subsequent delayed (24-120 hour) time period, irrespective of actual response in the delayed phase. However, participants who vomited or retched or received rescue medication in the delayed (24-120 hours) phase were not considered as failures in the acute (0-24 hours) phase. The overall phase began at the start of the administration of the oxaliplatin infusion. Percentage of participants who achieved a complete response in the overall phase of Cycle 2 are presented.
Time Frame: 0 to 120 hours in the second cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants | 84 | 90
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg; Test type: Superiority or Other; p = 0.0317, Pooled Z test — p-value based on normal approximation to the binomial using a pooled Z test; Treatment difference (%) = 6.0, 95% CI 2-sided [0.5 to 11.5]

5. Secondary Outcome: Maximum Nausea Score, Assessed by a Visual Analogue Scale (VAS)
Description: VAS was used to assess severity of nausea. The participants rated the severity of nausea by marking a line on a 100 millimeter (mm) (0 to 100 mm) long scale. A line placed on the extreme left, that is 0 mm indicated no nausea and extreme right that is 100 mm indicated nausea as bad as it can be. This scale has no subscales. The participant perception of their symptoms was measured using the VAS.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Scores on a Scale
  0-120 hours: number analyzed (Participants) | 349 | 353
  0-120 hours | 13.5 (23.3) | 16.0 (24.5)
  0-24 hours: number analyzed (Participants) | 286 | 288
  0-24 hours | 4.3 (12.9) | 5.3 (13.3)
  24-120 hours: number analyzed (Participants) | 349 | 352
  24-120 hours | 13.0 (22.6) | 15.3 (24.2)
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.0560, Wilcoxon-rank sum test
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.0443, Wilcoxon-rank sum test
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.1709, Wilcoxon-rank sum test

6. Secondary Outcome: Percentage of Participants Who Received Rescue Medication
Description: Anti-emetic rescue medication was defined as medication that was administered specifically for the treatment of nausea and/or emesis during Days 1-6 of each cycle. The choice of rescue anti-emetic medication was left to the discretion of the investigator. Participants who required antiemetic rescue medication(s) during the 120-hour assessment period were considered treatment failures for that cycle. Percentage of participants who received rescue medication are presented.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  0-120 hours | 9 | 8
  0-24 hours | 2 | 1
  24-120 hours | 9 | 8
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.3986, Chi-squared; Treatment difference (%) = -1.8, 95% CI 2-sided [-5.9 to 2.3]
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.3545, Chi-squared; Treatment difference (%) = -0.9, 95% CI 2-sided [-2.7 to 1.0]
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.3986, Chi-squared; Treatment difference (%) = -1.8, 95% CI 2-sided [-5.9 to 2.3]

7. Secondary Outcome: Percentage of Participants Who Vomited and/or Retched
Description: Vomiting was defined as the forceful expulsion of gastrointestinal contents through the mouth or nose. Retching was defined as the labored, spasmodic, rhythmic contraction of the respiratory and abdominal muscles in an attempt to vomit, that is not productive of gastrointestinal contents (also known as dry heaves). If a participant took rescue medication but there was no evidence of vomiting or retching, then the participant was considered as not having vomited. Percentage of participants who vomited and/or retched during the first 120 hours of the first cycle of chemotherapy are presented.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  0-120 hours | 11 | 10
  0-24 hours | 3 | 2
  24-120 hours | 11 | 10
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.6795, Chi-squared; Treament Difference (%) = -0.9, 95% CI 2-sided [-5.4 to 3.5]
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.4507, Chi-squared; Treament Difference (%) = -0.9, 95% CI 2-sided [-3.1 to 1.4]
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.6795, Chi-squared; Treament Difference (%) = -0.9, 95% CI 2-sided [-5.4 to 3.5]

8. Secondary Outcome: Percentage of Participants Who Reported Significant Nausea, Defined as a Maximum Score >= 25 mm on the VAS
Description: VAS was used to assess severity of nausea. The participants rated the severity of nausea by marking a line on a 100 mm (0 to 100 mm) long scale. A line placed on the extreme left, that is 0 mm indicated no nausea and extreme right that is 100 mm indicated nausea as bad as it can be. This scale has no subscales. The participant perception of their symptoms was measured using the VAS. Percentage of participants who reported significant nausea, defined as a maximum score >= 25 mm on the VAS are presented.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  0-120 hours | 19 | 21
  0-24 hours | 4 | 5
  24-120 hours | 19 | 21
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.4846, Chi-squared; Difference in percentage of participants = 2.1, 95% CI 2-sided [-3.8 to 8.0] — Difference in percentage of participants with response
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.6101, Chi-squared; Difference in percentage of participants = 0.8, 95% CI 2-sided [-2.3 to 3.9] — Difference in percentage of participants with response
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.4846, Chi-squared; Percentage of participants = 2.1, 95% CI 2-sided [-3.8 to 8.0] — Difference in percentage of participants with response

9. Secondary Outcome: Percentage of Participants Who Reported Nausea, Defined as a Maximum Score of >= 5 mm on the VAS
Description: VAS was used to assess severity of nausea. The participants rated the severity of nausea by marking a line on a 100 mm (0 to 100 mm) long scale. A line placed on the extreme left, that is 0 mm indicated no nausea and extreme right that is 100 mm indicated nausea as bad as it can be. This scale has no subscales. The participant perception of their symptoms was measured using the VAS. Percentage of participants who reported nausea, defined as a maximum score of >= 5 mm on the VAS are presented.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  0-120 hours | 37 | 45
  0-24 hours | 12 | 15
  24-120 hours | 37 | 45
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.1356, Chi-squared; Difference in percentage of participants = 3.8, 95% CI 2-sided [-1.2 to 8.9] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.0280, Chi-squared; Difference in percentage of participants = 8.1, 95% CI 2-sided [0.9 to 15.4] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.0280, Chi-squared; Difference in percentage of participants = 8.1, 95% CI 2-sided [0.9 to 15.4] — The parameter estimated was difference in percentage of participants with response

10. Secondary Outcome: Percentage of Participants Who Achieved Complete Protection Defined as Complete Responders With no Significant Nausea
Description: Complete protection was defined as no vomiting/retching, no use of rescue medication and no significant nausea. Percentage of participants who achieved complete protection or complete responders with no significant nausea are presented.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  0-120 hours | 75 | 74
  0-24 hours | 93 | 93
  24-120 hours | 75 | 74
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.7799, Chi-squared; Difference in percentage of participants = -0.9, 95% CI 2-sided [-7.3 to 5.5] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.7883, Chi-squared; Difference in percentage of participants = 0.5, 95% CI 2-sided [-3.2 to 4.2] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.7799, Chi-squared; Difference in percentage of participants = -0.9, 95% CI 2-sided [-7.3 to 5.5] — The parameter estimated was difference in percentage of participants with response

11. Secondary Outcome: Percentage of Participants Who Achieved Total Control, Defined as Complete Responders Who Had no Nausea
Description: Total control was defined as no vomiting/retching, no use of rescue medication and no nausea. Percentage of participants who achieved total control or complete responders with no nausea are presented.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  0-120 hours | 61 | 54
  0-24 hours | 88 | 83
  24-120 hours | 61 | 54
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-120 hours); Test type: Superiority or Other; p = 0.0507, Chi-squared; Difference in percentage of participants = -7.3, 95% CI 2-sided [-15 to 0.0] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (0-24 hours); Test type: Superiority or Other; p = 0.0800, Chi-squared; Difference in percentage of participants = -4.7, 95% CI 2-sided [-9.9 to 0.5] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs Casopitant 90 mg (24-120 hours); Test type: Superiority or Other; p = 0.0507, Chi-squared; Difference in percentage of participants = -7.3, 95% CI 2-sided [-15 to 0.0] — The parameter estimated was difference in percentage of participants with response

12. Secondary Outcome: Percentage of Participants Whose Daily Life Activities Were Impacted in the Overall Phase of Cycle 1, Assessed by Functional Living Index-Emesis (FLIE) Questionnaire
Description: FLIE questionnaire specifically addresses the impact of nausea and vomiting on daily activities (physical, social and emotional function, ability to enjoy meals). It consists of 18 items with questions divided into two domains: Nausea (questions 1-9) and Vomiting (questions 10-18). Each item is scored on a VAS with 7 hatch marks. The scale is anchored at 1 (Not at all) and 7 (A great deal). For questions 1,2,4,5,7,8-10,12-14,16 and 17 the final score was calculated by subtracting the initial score from 100 for questions 3,6,11,15 and 18 the final score was the one provided in the dataset. The score for the nausea domain: ([sum of nausea item scores] ÷ [Number of items answered] x 9) and for vomiting domain: ([sum of vomiting item scores] ÷ [Number of items answered] x 9). The total score was the sum of the nausea and vomiting domain scores. Higher scores indicate less impairment on daily life as a result of nausea or vomiting.
Time Frame: 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Percentage of participants
  Nausea impact | 21.3 | 23.7
  Vomiting impact | 12.5 | 11.5
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Nausea Impact: Placebo vs. Casopitant 90 mg; Cycle 1 (0-120 hours); Test type: Superiority or Other; Difference in percentage of participants = -2.6, 97.5% CI 2-sided [-9.9 to 4.7] — The parameter estimated was difference in percentage of participants with response
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Vomiting Impact: Placebo vs. Casopitant 90 mg; Cycle 1 (0-120 hours); Test type: Superiority or Other; Difference in percentage of participants = 0.7, 97.5% CI [-5.2 to 6.6] — The parameter estimated was difference in percentage of participants with response

13. Secondary Outcome: Severity of Nausea in the Overall, Acute, and Delayed Phases of Cycle 1 Assessed by a Categorical Scale
Description: Participants were asked to rate the level of nausea he/she experienced over the previous (24 hours for a period of 120 hours following the administration of MEC), by placing a vertical mark on a VAS. The severity of nausea and was calculated by using a 0 - 100 VAS where 0 = No Nausea and 100 = Nausea as bad as it can be. The categorical scale assessed the participants severity of his/her nausea using the following: mild: Queasiness/upset stomach that is manageable and minimally (if at all) affects daily activities, moderate: increased queasiness, sometimes with the feeling of having to vomit/throw up (but not vomiting), that has significant negative effect on the daily activities (for example, being unable to work, eat and drink, prepare food, care for children or others) and severe: feeling sick and vomiting or feeling like you are going to vomit, and unable to perform most daily activities. Higher scores indicated worst outcome.
Time Frame: 0 to 24 hours, 24 to 120 hours and 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Participants
  0-120 hours: None | 218 | 192
  0-120 hours: Mild | 73 | 97
  0-120 hours: Moderate | 49 | 54
  0-120 hours: Severe | 12 | 12
  0-24 hours: None | 313 | 299
  0-24 hours: Mild | 23 | 40
  0-24 hours: Moderate | 13 | 15
  0-24 hours: Severe | 3 | 1
  24-120 hours: None | 218 | 192
  24-120 hours: Mild | 73 | 97
  24-120 hours: Moderate | 49 | 54
  24-120 hours: Severe | 12 | 12
Statistical Analysis 1: Comparison: Placebo vs Casopitant 90 mg; Placebo vs. Casopitant 90 mg: (0-120 hours) in Cycle 1; Test type: Superiority or Other; p = 0.1572, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Casopitant 90 mg; Placebo vs. Casopitant 90 mg: (0-24 hours) in Cycle 1; Test type: Superiority or Other; p = 0.2908, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Casopitant 90 mg; Placebo vs. Casopitant 90 mg: (24-120 hours) in Cycle 1; Test type: Superiority or Other; p = 0.1572, Chi-squared

14. Secondary Outcome: Single-dose Pharmacokinetic (PK) Parameters: Area Under the Curve (AUC) 0 to Infinity (0-∞), AUC 0 to t (0-t) and AUC 0 to 24 Hours (0-24) for Casopitant; AUC (0-t) and AUC (0-24) for Metabolites GSK525060, GSK517142 and GSK631832
Description: Blood samples were obtained during Cycle 1 at the following times relative to the investigational product administration: pre-dose, end of infusion, 0.5, 1, 3, 5, 8, 12, 16, and 24 hours after the end of infusion. A final PK sample was collected between 30 and 48 hours after the investigational product infusion had completed. The actual time each sample was collected was captured to the nearest minute in the electronic case report form (eCRF). Following unblinding, only those participants who had been randomized to receive casopitant were included in the PK analyses. AUC(0-∞), AUC(0-t), AUC(0-24) for casopitant and metabolites GSK525060, GSK517142 and GSK631832 are presented.
Time Frame: Pre-dose, end of infusion and 0.5, 1, 3, 5, 8, 12, 16, 24 hours after the end of infusion
Population: PK parameter population: All participants who consented to PK sampling, who were randomized to IV casopitant and for whom a PK sample was obtained and analyzed, and from whom sufficient data was available to calculate casopitant PK parameters on an as-treated basis. Only those participants with data available at indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/milliliter (hr*ng/mL)
Arm/Group | Casopitant 90 mg
Number analyzed (Participants) | 29
Hour*nanogram/milliliter (hr*ng/mL)
  Casopitant: AUC(0-24) | 6913.626 (61.4868)
  Casopitant: AUC(0-inf): number analyzed (Participants) | 28
  Casopitant: AUC(0-inf) | 8607.049 (61.8698)
  Casopitant: AUC(0-t) | 7688.562 (58.9620)
  GSK525060: AUC(0-24) | 2247.290 (36.6378)
  GSK525060: AUC(0-t) | 2796.734 (36.6862)
  GSK517142: AUC(0-24): number analyzed (Participants) | 24
  GSK517142: AUC(0-24) | 49.964 (40.5170)
  GSK517142: AUC(0-t): number analyzed (Participants) | 26
  GSK517142: AUC(0-t) | 40.997 (126.8389)
  GSK631832: AUC(0-24) | 165.550 (38.6564)
  GSK631832: AUC(0-t) | 231.018 (40.8915)

15. Secondary Outcome: Single-dose Pharmacokinetic Parameters: Maximum Observed Drug Concentration (Cmax) for Casopitant and Metabolites GSK525060, GSK517142 and GSK631832
Description: Blood samples were obtained during Cycle 1 at the following times relative to the investigational product administration: pre-dose, end of infusion, 0.5, 1, 3, 5, 8, 12, 16, and 24 hours after the end of infusion. A final PK sample was collected between 30 and 48 hours after the investigational product infusion had completed. The actual time each sample was collected was captured to the nearest minute in the electronic case report form (eCRF). Following unblinding, only those participants who had been randomized to receive casopitant were included in the PK analyses. (Cmax) for casopitant and metabolites GSK525060, GSK517142 and GSK631832 are presented.
Time Frame: Pre-dose, end of infusion and 0.5, 1, 3, 5, 8, 12, 16, 24 hours after the end of infusion
Population: PK Parameter population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Casopitant 90 mg
Number analyzed (Participants) | 29
Nanogram/milliliter (ng/mL)
  Casopitant | 2078.776 (144.8121)
  GSK525060 | 143.038 (32.7047)
  GSK517142: number analyzed (Participants) | 28
  GSK517142 | 3.426 (45.1672)
  GSK631832 | 9.853 (35.8595)

16. Secondary Outcome: Single-dose Pharmacokinetic Parameters: Time to Maximum Observed Drug Concentration (Tmax) and Observed Elimination Half-life (t1/2) for Casopitant and Metabolites GSK525060, GSK517142 and GSK631832
Description: Blood samples were obtained during Cycle 1 at the following times relative to the investigational product administration: pre-dose, end of infusion, 0.5, 1, 3, 5, 8, 12, 16, and 24 hours after the end of infusion. A final PK sample was collected between 30 and 48 hours after the investigational product infusion had completed. The actual time each sample was collected was captured to the nearest minute in the eCRF. Following unblinding, only those participants who had been randomized to receive casopitant were included in the PK analyses. Tmax and t1/2 for casopitant and metabolites GSK525060, GSK517142 and GSK631832 are presented.
Time Frame: Pre-dose, end of infusion and 0.5, 1, 3, 5, 8, 12, 16, 24 hours after the end of infusion
Population: PK parameter population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Casopitant 90 mg
Number analyzed (Participants) | 29
Hour
  Casopitant: Tmax | 0.520 [0.00 to 1.50]
  Casopitant: t1/2: number analyzed (Participants) | 28
  Casopitant: t1/2 | 12.347 [5.68 to 28.76]
  GSK525060: Tmax | 3.580 [1.00 to 24.50]
  GSK517142: Tmax: number analyzed (Participants) | 28
  GSK517142: Tmax | 1.500 [0.58 to 24.50]
  GSK631832: Tmax | 5.500 [3.48 to 24.67]

17. Secondary Outcome: Single-dose Pharmacokinetic Parameters: Clearance (CL) for Casopitant
Description: Blood samples were obtained during Cycle 1 at the following times relative to the investigational product administration: pre-dose, end of infusion, 0.5, 1, 3, 5, 8, 12, 16, and 24 hours after the end of infusion. A final PK sample was collected between 30 and 48 hours after the investigational product infusion had completed. The actual time each sample was collected was captured to the nearest minute in the eCRF. Following unblinding, only those participants who had been randomized to receive casopitant were included in the PK analyses. CL for casopitant is presented.
Time Frame: Pre-dose, end of infusion and 0.5, 1, 3, 5, 8, 12, 16, 24 hours after the end of infusion
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Casopitant 90 mg
Number analyzed (Participants) | 28
Liter/hour | 10.457 (61.8700)

18. Secondary Outcome: Single-dose Pharmacokinetic Parameters: Volume of Distribution (Vdss) for Casopitant
Description: Blood samples were obtained during Cycle 1 at the following times relative to the investigational product administration: pre-dose, end of infusion, 0.5, 1, 3, 5, 8, 12, 16, and 24 hours after the end of infusion. A final PK sample was collected between 30 and 48 hours after the investigational product infusion had completed. The actual time each sample was collected was captured to the nearest minute in the eCRF. Following unblinding, only those participants who had been randomized to receive casopitant were included in the PK analyses. Vdss for casopitant is presented.
Time Frame: Pre-dose, end of infusion and 0.5, 1, 3, 5, 8, 12, 16, 24 hours after the end of infusion
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Casopitant 90 mg
Number analyzed (Participants) | 28
Liter | 126.776 (95.6229)

19. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly or birth defect. Any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product was recorded from the time a participant consents to participate in the study up to and including any follow-up contact.
Time Frame: Up to 35 days
Population: Safety Population which comprised of all participants who were randomized, and received any investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Participants
  AE | 176 | 171
  SAE | 23 | 26

20. Secondary Outcome: Number of Participants With Hematology Toxicity Grade Shifts From Baseline to Toxicity Grade 3 and 4
Description: Grade shifts from Baseline were assessed as shift from any Grade to Grade 3 or Grade 4 in any cycle. Toxicities were graded according to the National Cancer Institute common toxicity criteria for adverse events (NCI-CTCAE), version 3.0. Grade refers to the severity of the toxicity. The NCI-CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on the following general guideline: Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE and Grade 5: Death related to AE. It was assessed on Baseline (Day 1), during Day 6-10 and end of cycle. Hematology parameters assessed were hematocrit, hemoglobin, platelet count, total neutrophils and white blood cell count. Data has been presented for the number of participants with hematology toxicity grade shifts from Baseline to toxicity grade 3 and 4 for all cycles in a consolidated format.
Time Frame: Baseline (Day 1) to Day 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Participants
  Hematocrit: All cycles, Grade 2 to Grade 3 | 0 | 1
  Hemoglobin: All cycles, Grade 1 to Grade 3 | 2 | 0
  Hemoglobin: All cycles, Grade 2 to Grade 3 | 3 | 1
  Hemoglobin: All cycles, Grade 3 to Grade 3 | 0 | 2
  Platelet count: All cycles, Grade 0 to 3 | 1 | 1
  Total Neutrophils: All cycles, Grade 0 to 3 | 24 | 37
  Total Neutrophils: All cycles, Grade 1 to 3 | 0 | 1
  Total Neutrophils: All cycles, Grade 2 to 3 | 1 | 0
  White Blood Cell count: All cycles, Grade 0 to 3 | 10 | 5
  White Blood Cell count: All cycles, Grade 1 to 3 | 0 | 1
  White Blood Cell count: All cycles, Grade 2 to 3 | 1 | 2

21. Secondary Outcome: Number of Participants With Clinical Chemistry Toxicity Grade Shifts From Baseline to Toxicity Grade 3 and 4
Description: Grade shifts from Baseline were assessed as shift from any Grade to Grade 3 or Grade 4 in any cycle. Toxicities were graded according to the NCI-CTCAE, version 3.0. Grade refers to the severity of the toxicity. The NCI-CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on the following general guideline: Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE and Grade 5: Death related to AE. It was assessed on Baseline (Day 1), during Day 6-10 and end of cycle. Clinical chemistry parameters assessed were alanine amino transferase (ALT), aspartate amino transferase (AST), chloride, glucose, potassium, sodium and total bilirubin. Data has been presented for the number of participants with chemistry toxicity grade shifts from Baseline to toxicity grade 3 and 4 for all cycles in a consolidated format.
Time Frame: Up to Day 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Participants
  ALT: All cycles, Grade 0 to 3 | 1 | 2
  ALT: All cycles, Grade 2 to 3 | 1 | 0
  AST: All cycles, Grade 0 to 3 | 0 | 1
  High chloride: All cycles, Grade 1 to 3 | 2 | 0
  Low chloride: All cycles, Grade 0 to 3 | 0 | 1
  Hyperglycemia: Al cycles, Grade 0 to 3 | 1 | 3
  Hyperglycemia: All cycles, Grade 1 to 3 | 1 | 2
  Hyperglycemia: All cycles, Grade 2 to 3 | 9 | 5
  Hyperglycemia: All cycles, Grade 3 to 3 | 3 | 3
  Hypoglycemia: All cycles, Grade 0 to 4 | 1 | 1
  Hyperkalemia: All cycles, Grade 2 to 3 | 1 | 0
  Hyperkalemia: All cycles, Grade 4 to 3 | 1 | 0
  Hyperkalemia: All cycles, Grade 0 to 3 | 0 | 2
  Hyperkalemia: All cycles, Grade 0 to 4 | 0 | 2
  Hypokalemia: All cycles, Grade 0 to 3 | 6 | 8
  Hyponatremia: All cycles, Grade 1 to 3 | 6 | 8
  Total Bilirubin: All cycles, Grade 0 to 3 | 1 | 1
  Total Bilirubin: All cycles, Grade 0 to 4 | 1 | 0

22. Secondary Outcome: Evaluation of Vital Signs: Mean Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Vital signs assessment included DBP and SBP. SBP and DBP were recorded at Screening, on Day 1 of each cycle immediately before start of the investigational product infusion, at the completion of the infusion, and immediately after the end of the oxaliplatin infusion, then again at each end of cycle visit. Mean SBP and DBP are presented.
Time Frame: Up to End of Cycle for 6 cycles, an average of 24 days per cycle
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Millimeters of mercury (mmHg)
  DBP: Cycle 1, post-oxaliplatin: number analyzed (Participants) | 337 | 349
  DBP: Cycle 1, post-oxaliplatin | 77.2 (8.21) | 76.5 (8.27)
  DBP: Cycle 1, End of cycle: number analyzed (Participants) | 344 | 349
  DBP: Cycle 1, End of cycle | 76.9 (9.34) | 76.5 (9.80)
  DBP: Cycle 2, post-oxaliplatin: number analyzed (Participants) | 317 | 328
  DBP: Cycle 2, post-oxaliplatin | 77.7 (8.83) | 76.8 (8.86)
  DBP: Cycle 2, End of cycle: number analyzed (Participants) | 318 | 327
  DBP: Cycle 2, End of cycle | 76.8 (9.01) | 77.1 (9.89)
  DBP: Cycle 3, post-oxaliplatin: number analyzed (Participants) | 283 | 291
  DBP: Cycle 3, post-oxaliplatin | 78.0 (9.57) | 76.6 (9.25)
  DBP: Cycle 3, End of cycle: number analyzed (Participants) | 285 | 294
  DBP: Cycle 3, End of cycle | 77.3 (8.64) | 77.2 (9.80)
  DBP: Cycle 4, post-oxaliplatin: number analyzed (Participants) | 258 | 269
  DBP: Cycle 4, post-oxaliplatin | 78.2 (8.98) | 76.9 (9.16)
  DBP: Cycle 4, End of cycle: number analyzed (Participants) | 262 | 266
  DBP: Cycle 4, End of cycle | 76.8 (8.41) | 76.4 (9.90)
  DBP: Cycle 5, post-oxaliplatin: number analyzed (Participants) | 224 | 245
  DBP: Cycle 5, post-oxaliplatin | 77.4 (8.44) | 77.7 (9.55)
  DBP: Cycle 5, End of cycle: number analyzed (Participants) | 232 | 247
  DBP: Cycle 5, End of cycle | 77.1 (8.03) | 77.7 (9.84)
  DBP: Cycle 6, post-oxaliplatin: number analyzed (Participants) | 207 | 226
  DBP: Cycle 6, post-oxaliplatin | 77.9 (8.28) | 77.6 (9.01)
  DBP: Cycle 6, End of cycle: number analyzed (Participants) | 213 | 227
  DBP: Cycle 6, End of cycle | 77.9 (8.36) | 77.5 (8.83)
  SBP: Cycle 1, post-oxaliplatin: number analyzed (Participants) | 337 | 349
  SBP: Cycle 1, post-oxaliplatin | 130.6 (15.61) | 126.8 (14.11)
  SBP: Cycle 1, End of cycle: number analyzed (Participants) | 344 | 349
  SBP: Cycle 1, End of cycle | 128.7 (16.49) | 126.7 (15.04)
  SBP: Cycle 2, post-oxaliplatin: number analyzed (Participants) | 317 | 328
  SBP: Cycle 2, post-oxaliplatin | 130.1 (15.94) | 129.3 (15.61)
  SBP: Cycle 2, End of cycle: number analyzed (Participants) | 318 | 327
  SBP: Cycle 2, End of cycle | 128.9 (14.93) | 127.8 (15.30)
  SBP: Cycle 3, post-oxaliplatin: number analyzed (Participants) | 283 | 291
  SBP: Cycle 3, post-oxaliplatin | 131.0 (17.00) | 128.7 (15.57)
  SBP: Cycle 3, End of cycle: number analyzed (Participants) | 285 | 294
  SBP: Cycle 3, End of cycle | 128.8 (15.17) | 127.7 (15.58)
  SBP: Cycle 4, post-oxaliplatin: number analyzed (Participants) | 258 | 269
  SBP: Cycle 4, post-oxaliplatin | 131.8 (16.37) | 129.0 (15.96)
  SBP: Cycle 4, End of cycle: number analyzed (Participants) | 262 | 266
  SBP: Cycle 4, End of cycle | 128.0 (14.06) | 128.3 (15.39)
  SBP: Cycle 5, post-oxaliplatin: number analyzed (Participants) | 224 | 245
  SBP: Cycle 5, post-oxaliplatin | 131.3 (16.53) | 129.7 (16.01)
  SBP: Cycle 5, End of cycle: number analyzed (Participants) | 232 | 247
  SBP: Cycle 5, End of cycle | 128.6 (15.43) | 128.8 (15.82)
  SBP: Cycle 6, post-oxaliplatin: number analyzed (Participants) | 207 | 226
  SBP: Cycle 6, post-oxaliplatin | 132.2 (15.61) | 131.5 (17.07)
  SBP: Cycle 6, End of cycle: number analyzed (Participants) | 213 | 227
  SBP: Cycle 6, End of cycle | 129.7 (14.65) | 129.1 (15.04)

23. Secondary Outcome: Evaluation of Vital Signs: Mean Heart Rate
Description: Vital sign included heart rate which was recorded at Screening, on Day 1 of each cycle immediately before start of the investigational product infusion, at the completion of the infusion, and immediately after the end of the oxaliplatin infusion, then again at each end of cycle visit. Mean heart rate is presented.
Time Frame: Up to End of Cycle for 6 cycles, an average of 24 days per cycle
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Beats/minute
  Cycle 1, post-oxaliplatin: number analyzed (Participants) | 337 | 347
  Cycle 1, post-oxaliplatin | 73.1 (8.90) | 73.7 (9.45)
  Cycle 1, End of cycle: number analyzed (Participants) | 343 | 349
  Cycle 1, End of cycle | 75.1 (9.65) | 75.3 (9.91)
  Cycle 2, post-oxaliplatin: number analyzed (Participants) | 317 | 328
  Cycle 2, post-oxaliplatin | 73.0 (9.24) | 73.7 (9.39)
  Cycle 2, End of cycle: number analyzed (Participants) | 318 | 327
  Cycle 2, End of cycle | 74.8 (9.48) | 74.7 (9.79)
  Cycle 3, post-oxaliplatin: number analyzed (Participants) | 282 | 292
  Cycle 3, post-oxaliplatin | 73.2 (9.37) | 72.2 (9.16)
  Cycle 3, End of cycle: number analyzed (Participants) | 285 | 294
  Cycle 3, End of cycle | 74.9 (9.24) | 75.4 (10.56)
  Cycle 4, post-oxaliplatin: number analyzed (Participants) | 257 | 269
  Cycle 4, post-oxaliplatin | 72.6 (9.32) | 72.2 (9.16)
  Cycle 4, End of cycle: number analyzed (Participants) | 262 | 266
  Cycle 4, End of cycle | 75.0 (10.02) | 74.7 (9.36)
  Cycle 5, post-oxaliplatin: number analyzed (Participants) | 224 | 244
  Cycle 5, post-oxaliplatin | 72.8 (9.27) | 72.9 (9.35)
  Cycle 5, End of cycle: number analyzed (Participants) | 232 | 247
  Cycle 5, End of cycle | 74.7 (10.29) | 75.0 (9.10)
  Cycle 6, post-oxaliplatin: number analyzed (Participants) | 207 | 226
  Cycle 6, post-oxaliplatin | 73.5 (9.44) | 73.4 (9.72)
  Cycle 6, End of cycle: number analyzed (Participants) | 213 | 227
  Cycle 6, End of cycle | 74.7 (8.52) | 75.6 (10.22)

24. Secondary Outcome: Time to First Anti-emetic Rescue Medication
Description: Time to first rescue medication was defined as the length of time from initiation of oxaliplatin till the first reported use of a rescue medication. Participants withdrawing prematurely during the 120 hour assessment period without having received a rescue medication were assumed to have done so and the time of rescue medication was set to 0 hours. The first quartile for time to use of anti-emetic rescue medication was evaluated when 25th percentile of participants of MITT population reported use of anti-emetic rescue medication. Similarly, median and 75th percentile of participants of MITT population was planned to be reported. If, less than 25th percentile of participants reported use of anti-emetic rescue medication at the end of the 120 hour time period, then the observation was censored for the purpose of this analysis and in such case the data was planned to be reported as not evaluable (NA).
Time Frame: 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Hours | NA [NA to NA] — NA indicates 'median is not evaluable' as less than 25th percentile of participants reported use of anti-emetic rescue medication. | NA [NA to NA] — NA indicates 'median is not evaluable' as less than 25th percentile of participants reported use of anti-emetic rescue medication.

25. Secondary Outcome: Time to First Emetic Event
Description: Time to first emetic event was defined as the length of time from initiation of oxaliplatin until the time of first emetic event. Participants withdrawing prematurely from the study without having experienced an emetic event were assumed to have done so and the time of emetic event was set to 0 hours. The first quartile for time to emetic event was evaluated when 25th percentile of participants of MITT population reported emetic event. Similarly, median and 75th percentile of participants of MITT population was planned to be reported. If, less than 25th percentile of participants reported emetic event at the end of the 120 hour time period, then the observation was censored for the purpose of this analysis and in such case the data was planned to be reported as not evaluable (NA).
Time Frame: 0 to 120 hours in the first cycle of chemotherapy
Population: MITT Population.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Placebo | Casopitant 90 mg
Number analyzed (Participants) | 352 | 355
Hours | NA [NA to NA] — NA indicates 'median is not evaluable' as less than 25th percentile of participants reported emetic event. | NA [NA to NA] — NA indicates 'median is not evaluable' as less than 25th percentile of participants reported emetic event.

ADVERSE EVENTS:
Time Frame: Up to 35 days.
Description: SAE and non-SAE were collected and are reported for the Safety Population.
Arm/Group | Placebo | Casopitant 90 mg
All-Cause Mortality (participants affected / at risk) | 5/352 | 4/355
Serious Adverse Events (participants affected / at risk) | 23/352 | 26/355
Other Adverse Events (participants affected / at risk) | 237/352 | 257/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=352) | Casopitant 90 mg (N=355)
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=352) | Casopitant 90 mg (N=355)
Diarrhoea (Gastrointestinal disorders) | 74 | 96
Nausea (Gastrointestinal disorders) | 74 | 88
Constipation (Gastrointestinal disorders) | 39 | 38
Vomiting (Gastrointestinal disorders) | 35 | 16
Stomatitis (Gastrointestinal disorders) | 22 | 21
Dyspepsia (Gastrointestinal disorders) | 19 | 21
Abdominal pain (Gastrointestinal disorders) | 22 | 13
Neutropenia (Blood and lymphatic system disorders) | 94 | 108
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 38
Anaemia (Blood and lymphatic system disorders) | 26 | 14
Leukopenia (Blood and lymphatic system disorders) | 23 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 46
Paraesthesia (Nervous system disorders) | 36 | 24
Neuropathy peripheral (Nervous system disorders) | 29 | 30
Headache (Nervous system disorders) | 18 | 26
Fatigue (General disorders) | 56 | 53
Anorexia (Metabolism and nutrition disorders) | 30 | 24
Hypertension (Vascular disorders) | 15 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.